CLINICAL TRIAL: NCT00205296
Title: Effect of Fitness Training on Insulin Sensitivity and Body Composition in Children
Brief Title: Fitness Training in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-090
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2008-10

CONDITIONS: Obesity; Low Fitness
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: exercise — this will test the effect of exercise on insulin sensitivity, fitness and body composition

SUMMARY:
We hypothesize that improvement in cardiovascular fitness is associated with a greater improvement in insulin sensitivity than improvement in body composition (loss of body fat) is associated with insulin sensitivity. Towards that we are randomizing children who are overweight, or children with low fitness levels to exercise intervention 2 or three times per week.

ELIGIBILITY:
Inclusion Criteria:

* obesity
* low fitness

Exclusion Criteria:

* diagnosis of diabetes
* inability to exercise

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2002-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
maximal VO2 levels | 9 months

SECONDARY OUTCOMES:
fasting insulin and glucose levels | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Carrel, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States